CLINICAL TRIAL: NCT03405025
Title: Feasibility Study of RadioFrequency Endoscopic ABlation, With ULtrasound Guidance, as a Non-surgical, Adrenal Sparing Treatment for Aldosterone-producing Adenomas
Brief Title: Radiofrequency Endoscopic Ablation With Ultrasound Guidance: a Non-surgical Treatment for Aldosterone-producing Adenomas
Acronym: FABULAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Queen Mary University of London (Other); British Heart Foundation (Other); University of Cambridge (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 222446
Record Dates: First submitted 2017-12-21; First posted 2018-01-19 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Primary Hyperaldosteronism; Primary Hyperaldosteronism Due to Adrenal Adenoma
MeSH Terms: conditions — Hyperaldosteronism | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: All participants will undergo the intervention: endoscopic ultra-sound guided radiofrequency ablation of their left adrenal aldosterone producing adenoma. The primary outcome is safety and feasibility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety and Feasibility (Other): All patients will undergo endoscopic US guided radiofrequency ablation, to assess safety and feasibility.
  Interventions: Procedure: Endoscopic ultrasound guided radiofrequency ablation; Device: ultrasound

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided radiofrequency ablation — To establish if radiofreuqency ablation of aldosterone producing adrenal adenomas can be carried out via the endoscopic route and to assess safety of the procedure.
Device: ultrasound — ultrasound

SUMMARY:
High blood pressure (hypertension) causes strokes and heart attacks. While most patients need long-term treatment with pills, some have a cause which can be removed, curing the hypertension. The commonest curable cause is a benign nodule in one of the hormone glands, the adrenals. About one in 20 patients have such a nodule, but difficulties with diagnosis, and reluctance to proceed to surgery for a benign condition, limit the number having adrenal gland surgery to fewer than 300 per year in the UK. A potential, and exciting, solution to this dilemma is to use a momentary electric current to cauterise the nodule (radiofrequency ablation), without affecting the rest of the adrenal gland, and avoiding the need for surgery. Nodules in the left adrenal gland are easily reached under mild sedation using a similar procedure as is standard for investigating stomach ulcers (endoscopy). The study is designed to show that this approach (endoscopic ultrasound guided radiofrequency ablation) is very safe, and to provide initial evidence that the hormone abnormality is cured.

DETAILED DESCRIPTION:
Primary hyperaldosteronism (PA) is one of the commonest causes of hypertension. It is estimated to be the root cause in 10% of all patients with hypertension and 20% of all patients with resistant hypertension. Conventionally, patients with PA are divided 50:50 into those with a curable, unilateral aldosterone-producing adenoma (APA), and those with bilateral idiopathic adrenal hyperplasia (IAH).

Individual clinicians may reasonably consider it unnecessary to diagnose a benign condition whose work-up for surgery can be arduous, and the benefits uncertain. Public health doctors could reasonably despair at a large increase in demand for scarce surgical resources, when long term comparison of medical and surgical approaches have not been undertaken. Yet PA is regarded as a high-risk subset of hypertension, with an estimated 4-12 fold excess rate of cardiovascular complications compared to otherwise comparable patients with Hypertension. The American Endocrine Society Guidance recommends that where resources permit, a unilateral APA should be removed in order to protect patients from the long-term consequences of excess aldosterone. At present, most APAs are removed by key-hole surgery, with a 2% conversion rate to open surgery.

While such surgery is justified by the serious cardiovascular risk of PA, the high level of proof (of unilateral disease) before surgical referral has the paradoxical outcome of reducing take-up of a procedure that can be life-prolonging. A further paradox is that the rigid division of PA into unilateral adenoma vs bilateral hyperplasia is probably incorrect and that an intervention which does not require the distinction may, in stages, come to be regarded as the more logical approach to cure of PA, with reduction/prevention of cardiovascular risk. The obvious alternative intervention is selective ablation of APA(s), sparing most of the adjacent adrenal gland. Several publications report anecdotal success using this technique. The eligibility criteria for ablation were variable, but generally the patients were medically unfit or declined to undergo surgery. Success rates, measured as reversal of the biochemical abnormalities of PA, and radiological resolution, were high. However, there were few major adverse events. Most patients were monitored in hospital after the procedures, with shorter stays than the 2-3 days typical of most centres following laparoscopic surgery.

The investigators wish to progress from the experience with percutaneous and retroperitoneoscopic ablation to an approach which should maximise the ease and applicability of ablation whilst reducing the risk of adverse events. The primary outcome of the study will be safety. However, by the end of the study the investigators also need to have sufficient evidence of efficacy to justify, and guide design of, a subsequent multi-centre comparison trial.

Population Patients over the age of 18 diagnosed with left adrenal aldosterone producing adenoma meeting criteria from Endocrine Society clinical practice guidelines for primary hyperaldosteronism. The intervention (ultrasound guided endoscopic radiofrequency ablation) will be offered to those unsuitable for left adrenalectomy, who do not want surgery, or those who meet the criteria for surgery but wish to consent to radiofrequency ablation.

Design of study and intervention FABULAS is a three-center study, modelled on phase 1b/2a trials of novel drugs. It aims to determine the safety and efficacy study of endoscopic ultrasound-guided ablation as a nonsurgical, adrenal-sparing treatment for aldosterone-producing adenomas. Thirty patients will be enrolled onto the study comprised of three cohorts of ten patients. The three cohorts will run sequentially with overlapping stages, and the safety of the first six patients in each cohort/group will be reviewed before the next group commences.

Potential patients will be identified by referrals to our specialist Endocrine or Hypertension clinics. Once identified patients will be recruited at St. Bartholomew's Hospital in a Screening Visit where they will be clinically assessed, bloods and baseline investigations such as urinalysis and ECGs will be performed and informed consent gained for official enrolment onto the study.

Diagnostic PET CT scans using a tracer 11-C-Metomidate (or an alternative tracer, when available) will be used for confirmation of a left Conn's adenoma(s). Some patients may have already had this investigation as part of their work up. If so the PET CT does not need to be repeated. Group 1's (please see eligibility section for details) endoscopies will be managed in the Research Endoscopy Suite within the Clinical Research Facility at UCLH. Assuming group 1 is non-problematic, Barts Hospital will initiate ablations in year 2. The two-site approach maximises safety, assures recruitment of 1-2 eligible patients per month, and provides some early insight to the generalisability of the innovation.

Outcomes and assessment

The Primary Outcome Measures The primary outcome is safety, whether the recorded patient safety outcome data establishes that perforation, haemorrhage and infarction of major organs does not occur. This will be assessed at 48 hours.

This will be achieved by:

* Accurate adverse event reporting;
* Clinical assessment (history and examination) looking for features of blood loss, perforation, or inflammation/infarction of peri-adrenal tissues;
* Blood tests for Hb, WBC, and Renal function, amylase, LFTs, CRP; and.
* Urinalysis for blood and protein.

The Secondary Outcome Measures

The difference from baseline measurements at 3 and 6 months following ablation will be measured using the following clinical, biochemical and radiological parameters:

* Plasma electrolytes;,
* Aldosterone and renin ratio at 3 and 6 months;
* PET CT 3 months post ablation for radiological disappearance, diameter size and SUV measurements;.
* The reduced use or cessation of supplementary potassium medication; and
* Home BP (measured 3 readings twice a day for 4 days preceding clinic visit).Reduction in/or no longer taking antihypertensive medication

Assessment of cure will be performed at the site not involved in patient care. This will be subject to ratification by the safety committee who are not involved in the study.

Sample size / recruitment size A sample size of 30 patients will be recruited to the clinical trial. These statistical analyses have been performed by Dr Stephen Morant, University of Dundee (statistician). Patients will be identified through specialist endocrine / hypertension clinics and recruitment will be at St Bartholomew's Hospital.

The Intervention

Initially the patient's imaging (PET CT) will be reviewed at a multidisciplinary meeting to confirm the diagnosis and suitability for treatment by radiofrequency ablation for a left aldosterone producing adenoma. Currently this technique can only be used for the left adrenal gland due to its position near to the stomach.

On the day of the procedure the patient will receive a general anaesthetic or conscious sedation for the treatment. An endoscope with an ultrasound probe in the tip will be passed in to the stomach or small bowel to identify the adrenal adenoma.. A fine needle is then inserted into the adenoma via the endoscope and its contents aspirated. Samples will be sent to the laboratory for routine analysis. Following aspiration of the adenoma, the patient will undergo Endoscopic Ultrasound-Guided Radiofrequency Ablation (EUS-RFA) treatment. The radiofrequency probe will be placed into the adenoma via the needle. The needle will be withdrawn slightly so the probe lies within the adenoma. A low power current of 10 Watts for 90 seconds will then be applied to the lesion on up to 10 occasions to ablate the tumour. It is anticipated the treatment will cause destruction of the adenoma.

The 30 patients recruited to this study, will need to stay in hospital for approximately 48 hours following treatment. A CT scan will be performed 24-48 hours post ablation. Based on the experience so far, it is hoped that the side effects of radiofrequency ablation will be minor and that ultimately the treatment will be performed as a day-case procedure. If our initial experience confirms this, patients recruited to this study may be discharged on the same day as treatment, following review by the medical team. Patients will be followed up at one, three and six months in outpatients to recheck blood pressure and blood tests to check if the treatment has been successful, with a repeat PET CT scan prior to the appointment. Blood tests will also be performed on the day of the appointment, as part of standard care. If the adenoma has not been completely ablated at 3 months the patient may be offered a further EUS-RFA treatment.

Patients will be asked to measure their blood pressure at home 4 days before each study visit with a monitor loaned to them whilst on the clinical trial. In addition to formally checking for any adverse effects at each clinic visit, patients were also asked to report any side-effects encountered to the medical team.

Sample management Cytology from the fine needle aspiration will be sent for immunohistochemistry staining. RNA will be obtained to look expression of the enzymes that produce aldosterone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and above
2. Diagnosis of PHA based on published Endocrine Society guidelines
3. Positive serum aldosterone renin ratio (ARR) with another local diagnostic confirmatory test (MRI or CT imaging)

There are 3 inclusion subset groups:

Group 1

1. Left-sided APA proven on either AVS or PET CT.
2. Patients wishing to take fewer drugs for their hypertension.
3. Patients not usually referred for surgery because the benefit: risk is considered too low.
4. Patients aged ≥60 whose BP is at or near target (BP140/90 for most patient groups, BP 130/80 if co-morbidities listed in Hypertension guidelines) on treatment with four or more drugs.
5. patients with identified macroadenomas (APAs >= 1 cm in diameter), who have at least 1 cm of peri-adrenal fat on axial and coronal projections.

Group 2

Patients aged 18 years and above with diagnosis of PA and either:

[i] a definite unilateral left APA, but the patient does not want surgery; or [ii] probable but not unequivocal evidence of a unilateral left adrenal APA.

Group 3 Patients over 18 years of age meeting criteria for surgery, but consent to undergo endoscopic ablation instead.

Exclusion Criteria:

1. Inability to give informed consent.
2. Any patients continuing on beta blockers/direct renin blockers.
3. Pregnant women or those unable or unwilling to take secure contraceptive precautions.
4. Any illness, condition or drug regimen considered a contraindication by the PI/CI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events of endoscopic ultrasound-guided radiofrequency ablation. | 24-48 hours post procedure
  The primary objective is to test the primary hypothesis which states that endoscopic ultrasound-guided radiofrequency ablation of aldosterone-producing adenomas of the adrenal gland is a safe method for achieving sustained reduction in plasma aldosterone.
  Specifically this will be assess via number of patients in whom one of the following is reported:
  1. Major haemorrhage (seen on 24-48 hour safety CT)
  2. Fall in Hb
  3. Evidence of infarction of peri-adrenal organs on blood tests and CT
  4. Evidence of rupture of stomach on CT

SECONDARY OUTCOMES:
Evidence of 'biochemical cure' post endoscopic ultrasound-guided radiofrequency ablation | 6 months
  Difference in measurement of plasma electrolytes, renin and aldosterone at baseline and 6 months following ablation looking for normalisation post procedure. Definition of biochemical success defined as per PASO consensus
Evidence of 'radiological cure' post endoscopic ultrasound-guided radiofrequency ablation | 6 months
  Metomidate PET CT will be performed at 6 months after ablation and compared with baseline PET CT looking for 'radiological cure', ie successful ablation of previous 'hot' aldosterone producing adrenal adenoma.
Evidence of 'clinical cure' post endoscopic ultrasound-guided radiofrequency ablation | 6 months
  Difference in Home BP measurements (3 readings morning and 3 in the evening for 4 days) before clinic visits at baseline and at 6 months. Definition of clinical success defined as per PASO consensus. If home BP is not available, clinic BPs will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pereira, Principal Investigator — University College, London
Locations (3):
- United Kingdom (3):
  - University of Cambridge and Cambridge NIHR Biomedical Research Centre, Cambridge
  - Queen Mary University of London, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: Yes
Please see below
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol, SAP and ICF will be available within next 3-6 months and will remain available until close of study.
  The CSR will be available following statistical analysis.